CLINICAL TRIAL: NCT04658485
Title: The Modulatory Effect of Anodal Primary Motor Cortex and Cathodal Primary Somatosensory Cortex Transcranial Direct Current Stimulation on Pain Thresholds in the Neck Musculature.
Brief Title: The Effect of Transcranial Direct Current Stimulation of the Primary Motor and Somatosensory Cortex on Pain Thresholds.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aalborg University (Other)
Collaborators: Danish National Research Foundation (Other)
Responsible Party: Principal Investigator, Sebastian Kold Sørensen, PhD-fellow, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: N-20180085.p3
Record Dates: First submitted 2020-09-23; First posted 2020-12-08 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects are pseudo randomly allocated to either the active stimulation group or the sham stimulation group (placebo), ensuring equal weighting of male and female in the two groups. The care provider is handed the tDCS device which is preprogrammed by a third party either deliver the active or the sham stimulation based on the participation ID-number, effectively blinding the care provider. The outcome assessor and investigator is similarly blinded to the protocol administered to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator)
  Interventions: Device: Active tDCS
- Sham tDCS (Placebo Comparator)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Using the 2-channel neuro-stimulator Sooma tDCS equipment we provide 20 minutes of 2 mA anodal stimulation of the primary motor cortex (M1) with the cathode located over the right primary somatosensory cortex (S1).
  Arms: Active tDCS
Device: Sham tDCS — Using the 2-channel neuro-stimulator Sooma tDCS equipment we provide a sham stimulation with the anode place over the primary motor cortex (M1) and cathode located over the right primary somatosensory cortex (S1). The sham stimulation consists of 30 seconds of stimulation ramping up to a maximum of 2 mA, then 19 minutes of the device providing no stimulation and then ramping down from 2 mA intensity to 0 in the last 30 seconds. This configuration is designed to mimic the sensory experience of active tDCS.
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to investigate the modulatory effect of a novel tDCS configuration on the pain sensitivity in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the modulatory effect of a single session 20 min anodal primary motor cortex (M1) and cathodal primary somatosensory cortex (S1) transcranial direct current stimulation (tDCS) on the pain sensitivity on the descending part of musculus trapezius in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age between 18-30 years
* Living in Denmark

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Current use of opioids, antipsychotics, benzodiazepines
* Previous or current neurological, musculoskeletal, rheumatic, malignant, inflammatory or mental illnesses
* Current or prior chronic pain conditions
* Lack of ability to cooperate

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in pressure pain threshold | Two assessments total: Once before the stimulation intervention (baseline assessment) and once again three minutes after the stimulation (post intervention assessment).
  A hand-held pressure algometer (Somedic, Hörby, Sweden) with a 1-cm2 probe was used to record the pressure pain threshold. The pressure is increased gradually at a rate of 30 kPa/s. The measurement is repeated three times on descending part of the medial musculus trapezius sinister and dexter respectively.

SECONDARY OUTCOMES:
Change in Heat and Cold Pain Detection Thresholds | Two assessments total: Once before the stimulation intervention (baseline) and once again five minutes after the stimulation (post intervention assessment).
  A 3×3 cm (9 cm2) contact thermode (Medoc Advanced Medical Systems, Israel) was used to apply thermal stimulation. Each stimulus will be started at 32°C and thresholds of heat and cold pain detection was assessed by ascending or descending ramps in temperature to the cutoffs of 0-50 °C. This will be assessed on the skin over the left side descending part of the medial musculus trapezius.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Graven-Nielsen, Prof., Study Director — Aalborg University
Locations (1):
- Center for Neuroplasticity and Pain, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kold S, Kragh AJ, Graven-Nielsen CS, Elnegaard FS, Lund F, Vittrup IV, Cliff KL, Sivarooban R, Petrini L. Neuromodulation of somatosensory pain thresholds of the neck musculature using a novel transcranial direct current stimulation montage: a randomized double-blind, sham controlled study. Scand J Pain. 2022 Feb 7;22(3):622-630. doi: 10.1515/sjpain-2021-0187. Print 2022 Jul 26. PMID 35130374